CLINICAL TRIAL: NCT01038765
Title: Mindfulness Based Cognitive Therapy for Patients With Recurrent Depression: a Clinical Trial
Brief Title: Mindfulness Based Cognitive Therapy for Recurrent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Fonds Psychische Gezondheid (Other)
Responsible Party: Principal Investigator, Anne Speckens, Anne E.M. Speckens, Prof. dr., Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MFN-2005-2010; 2005 6028 (Other: Fonds Psychische Gezondheid, Netherlands (previously: NFGV))
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Depressive Disorder, Major
Keywords: Recurrent Major Depressive Disorder; Mindfulness Based Cognitive Therapy; Randomized Controlled Trial
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (Experimental): Mindfulness Based Cognitive Therapy
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Waiting list control group (No Intervention): 3-month waiting list group

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — 8-weeks group based intervention of mindfulness and cognitive behavioural techniques
  Other Names: MBCT
  Arms: Mindfulness Based Cognitive Therapy

SUMMARY:
The purpose of this study is to investigate the effectiveness and possible mediating factors of Mindfulness Based Cognitive Therapy (MBCT) for recurrent depression.

DETAILED DESCRIPTION:
Mindfulness Based Cognitive Therapy (MBCT) is a 8 session group intervention and is well described by several authors.

Previous studies showed Mindfulness Based Cognitive Therapy (MBCT) to be effective to prevent relapse in patients with recurrent depression and 3 or more previous depressive episodes.

Study aims are:

1. to replicate previous findings in The Netherlands, by a research team which did not develop the intervention
2. to investigate if MBCT is applicable for patients with recurrent depression and current depressive symptoms
3. to examine possible mediators of treatment effect and predictors of relapse in the year following the treatment

In this study, patients are randomly assigned to a MBCT intervention group or a waiting list control group. Patients allocated to the waiting list control condition will receive the MBCT course three months later. All patients who participated in a MBCT training will be assessed during the year following the completion of the MBCT course. We aim to include about 220 patients.

ELIGIBILITY:
Inclusion Criteria:

* 3 or more previous depressive episodes
* if treated with medication: constant dose of at least 6 weeks

Exclusion Criteria:

* Bipolar Disorder
* Psychotic disorder
* Neurological or somatic illness affecting depression or outcome measures
* Current alcohol or drugs dependency
* Acute need of psychiatric treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2005-01; Primary Completion 2010-03 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne EM Speckens, Prof. dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Background] Ma SH, Teasdale JD. Mindfulness-based cognitive therapy for depression: replication and exploration of differential relapse prevention effects. J Consult Clin Psychol. 2004 Feb;72(1):31-40. doi: 10.1037/0022-006X.72.1.31. PMID 14756612
- [Background] Barnhofer T, Crane C, Hargus E, Amarasinghe M, Winder R, Williams JM. Mindfulness-based cognitive therapy as a treatment for chronic depression: A preliminary study. Behav Res Ther. 2009 May;47(5):366-73. doi: 10.1016/j.brat.2009.01.019. Epub 2009 Feb 5. PMID 19249017
- [Background] Kenny MA, Williams JM. Treatment-resistant depressed patients show a good response to Mindfulness-based Cognitive Therapy. Behav Res Ther. 2007 Mar;45(3):617-25. doi: 10.1016/j.brat.2006.04.008. Epub 2006 Jun 23. PMID 16797486
- [Background] Kingston T, Dooley B, Bates A, Lawlor E, Malone K. Mindfulness-based cognitive therapy for residual depressive symptoms. Psychol Psychother. 2007 Jun;80(Pt 2):193-203. doi: 10.1348/147608306X116016. PMID 17535594
- [Derived] van Aalderen JR, Donders AR, Giommi F, Spinhoven P, Barendregt HP, Speckens AE. The efficacy of mindfulness-based cognitive therapy in recurrent depressed patients with and without a current depressive episode: a randomized controlled trial. Psychol Med. 2012 May;42(5):989-1001. doi: 10.1017/S0033291711002054. Epub 2011 Oct 3. PMID 22017808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were referred by their general practitioners or psychiatrists and psychologists in and around Nijmegen, the Netherlands. Alternatively, they were self-referred, informed by local and national advertisements.
Pre-assignment Details: Patients were excluded for not having three or more previous depressive episodes (N=19), change in medication within 6 weeks before the start of the study (N=4), previous (hypo)manic episodes (N=2), current substance abuse (N=3), acute need for psychiatric treatment (N=2), unsuitability for groups (N=2), cognitive impairments (N=1).
Groups:
- Mindfulness Based Cognitive Therapy: Mindfulness Based Cognitive Therapy
  Mindfulness Based Cognitive Therapy : 8-weeks group based intervention of mindfulness and cognitive behavioural techniques
- Waiting List Control Group (TAU): three month waiting list group receiving treatment as usual
Period: Overall Study
Arm/Group | Mindfulness Based Cognitive Therapy | Waiting List Control Group (TAU)
Started | 111 | 108
Completed | 102 | 103
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Waiting List Control Group (TAU): Three-month waiting list group receiving treatment as usual (TAU)
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Cognitive Therapy | Waiting List Control Group (TAU) | Total
Number analyzed (Participants) | 111 | 108 | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 111 | 108 | 219
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (11.5) | 47.7 (11.1) | 47.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 74 | 145
  Male | 40 | 34 | 74
Region of Enrollment [Number; unit: participants]
  Netherlands | 111 | 108 | 219

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms
Description: Hamilton Depression Rating Scale. The HAMD is a standardized 17-item interview to measure number and severity of depressive symptoms on a 0-52 score.
  Higher values indicate a worse outcome. Specifical, HAMD scores can be interpreted as "no depression" (0-7), "mild depression" (8-16), "moderate depression" (17-23) and "severe depression" (24-52).
Time Frame: Assessments were performed at 0, 3, 6, 9, 12, 15 months, and change between 3 and 0 months was the primary analysis.
Population: Due to missing values, 9 subjects in the MBCT group and 5 from the waiting list control group could not be analysed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Waiting List Control Group: Waiting list control group, from 0 to 3 months. Patients received usual care but not MBCT.
Arm/Group | Mindfulness Based Cognitive Therapy | Waiting List Control Group
Number analyzed (Participants) | 102 | 103
units on a scale | 7.5 (5.8) | 10.5 (6.8)

2. Secondary Outcome: Self-report Depressive Symptoms
Description: Beck Depression Inventory (BDI), a 21-item self-report questionnaire to measure depressive symptoms, score range 0-63.
  Higher scores indicate a worse outcome. Specifically, BDI scores can be interpreted as "minimal depression" (0-13), "mild depression" (14-19), "moderate depression" (20-28) and "severe depression" (29-63).
Time Frame: Assessments were performed at 0, 3, 6, 9, 12, 15 months, and change between 3 and 0 months was the primary analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Cognitive Therapy | Waiting List Control Group
Number analyzed (Participants) | 102 | 103
units on a scale | 10.3 (7.8) | 16.2 (9.8)

ADVERSE EVENTS:
Arm/Group | Mindfulness Based Cognitive Therapy | Waiting List Control Group (TAU)
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/108
Other Adverse Events (participants affected / at risk) | 0/111 | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes